CLINICAL TRIAL: NCT03921398
Title: Identifying New Therapeutic Targets for Lupus Treatment
Acronym: ELUDIAL
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: APHP180500
Record Dates: First submitted 2019-04-16; First posted 2019-04-19 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Lupus Nephritis
Keywords: Lupus nephritis; haemodialysis
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Blood and saliva samples Feces samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with ESRD: Patients with history of biopsy-proven lupus nephritis (all classes of lupus nephritis)
- Patients with active lupus prior to treatment and no ESRD: Patients with biopsy-proven ACTIVE lupus nephritis
- Healthy individuals: Healthy individuals

SUMMARY:
Lupus is an autoimmune disease affecting mainly young women (9/1). Lupus nephritis (LN) occurs in 30% of the cases of lupus and is associated with end stage renal disease (ESRD) in 17 to 25% of cases after 10 years. Overall, nearly 7% of lupus patients will develop ESRD due to LN. Historically, 5-year survival after LN was lower than 20%. Nowadays, 45% of patients suffer from multiple relapses that are associated with an intermediate risk of ESRD. When ESRD occurs, lupus activity decreases progressively to reach a stable extinct state. At this stage it is possible to stop all medications to control lupus, without any flare of lupus activity. Lupus extinction following ESRD corresponds to a state of complete remission. Obtaining such a result before ESRD would avoid damages to several organs and side effects of immunosuppressive therapy. Understanding the mechanisms responsible for lupus extinction following ESRD is an innovative approach to decipher lupus pathophysiology. The objective of the study is to identify the mechanisms responsible for lupus extinction and to propose new therapeutic options based on these new mechanisms. Mechanisms responsible for lupus extinction are unknown. Lupus extinction depends on the duration of ESRD. Accumulation of several toxins that kidneys would normally eliminate in the urine is a hallmark of ESRD. Such toxins are called "uremic toxins" since they accumulate during "uremia" (ESRD). They affect biological systems such as fertility and immunity that are both closely related to lupus pathophysiology. The investigators hypothesize that studying LN extinction after ESRD will provide novel therapeutic targets to extinct lupus before ESRD. To this end, they will investigate several non-exclusive hypotheses based on previous findings of our consortium, or issued from clinical observations: the sexual dysfunction hypothesis and the ESRD-associated immune cells dysfunction hypothesis. In parallel, they will conduct an open screening of new mechanisms underlying the lupus extinction through the characterization of the differential gene expression profile associated with lupus extinction in patients undergoing dialysis.

DETAILED DESCRIPTION:
Lupus is an autoimmune disease affecting mainly young women (9/1). Lupus nephritis (LN) occurs in 30% of patients and is associated with end stage renal disease (ESRD) in 17 to 25% of cases after 10 years. Overall, nearly 7% of lupus patients will develop ESRD due to LN. Historically, the 5-year survival after LN was below 20%. Nowadays, 45% of patients suffer from multiple relapses that are associated with an intermediate risk of ESRD. When ESRD occurs, lupus activity decreases progressively to reach a stable extinct state. At this stage it is possible to stop all medications to control lupus, without any flare of lupus activity. Lupus extinction following ESRD corresponds to a state of complete remission. Obtaining such a result before ESRD would prevent the damages of active lupus to several organs and side effects of immunosuppressive therapy. Understanding the mechanisms responsible for lupus extinction following ESRD is an innovative approach to decipher lupus pathophysiology.

The objective of this study is to identify the mechanisms responsible for lupus extinction in ESRD (candidate pathways) and to propose new therapeutic options targeting those candidates.

There is an important need for treatment innovation for systemic lupus and LN. A large number of biotherapies have been developed recently based on the known pathophysiology of the disease. Despite important efforts made by the medical community, many research groups, and pharmaceutical companies, randomized clinical trials (RCT) failed to validate innovative treatment strategies for several decades. This project proposes the identification of new treatment solutions through explorations in a field free of previous investigation in that aim.

A detailed knowledge of lupus extinction is required to understand its pathophysiology. This study will detail the timeframe of, and the factors associated with lupus extinction after ESRD. Moreover, previous investigations had been conducted separately in different projects and mainly provided descriptive results. Then a global and integrative strategy of research will be built in an attempt to embrace the subject as broadly as possible and maximize the opportunities to obtain successful outcome. The project will investigate specific hypotheses that were developed from the investigators' experience and based on the expertise of the consortium, both in lupus and immune dysfunction and in ESRD and uremic toxins. The addition of a "without a priori" approach by a systematic screening of gene expression associated with lupus extinction in haemodialysis will allow the investigators to propose a large panel of potential candidates to investigate further. Altogether, identifying the causes responsible for lupus extinction following ESRD is an innovative approach to discover new therapeutic targets. The investigators hypothesize that mimicking LN extinction due to ESRD provides a unique opportunity to propose new strategies to treat active lupus and LN before ESRD. The mechanisms responsible for lupus extinction are unknown. Lupus extinction depends on the duration of ESRD. Accumulation of several toxins that kidneys would normally eliminate in the urine is a hallmark of ESRD. Such toxins are called "uremic toxins" since they accumulate during "uremia" (ESRD). They affect biological systems such as fertility and immunity that are both closely related to lupus pathophysiology.

The investigators hypothesize that studying lupus extinction after ESRD will provide novel therapeutic targets to extinct lupus before ESRD. To this end, they propose to investigate several non-exclusive hypotheses based on previous findings: the sexual dysfunction hypothesis and the ESRD-associated immune cells dysfunction hypothesis. In parallel, they will conduct an open screening of new mechanisms underlying the lupus extinction through the characterization of the differential gene expression profile associated with lupus extinction in patients on chronic haemodialysis, comparing gene expression of dialysis patients with extinct lupus versus patients with still active lupus at the time of the study.

They first propose a comparison of active and extinct lupus in patients with ESRD. Lupus patients on chronic haemodialysis in Ile-de-France (n=75) will be recruited for the biological and clinical comparison between patients with persistent lupus activity to those with extinct lupus. These dialysis patients have been identified from the national REIN registry, which prospectively collects data for all incident patients undergoing renal replacement therapy (dialysis or kidney transplantation). A specific authorization was obtained from the Scientific Board of the REIN Registry at Agency of Biomedicine). Additionally, patients with active lupus prior to treatment and no ESRD will serve as a "positive control" group (n=45) for markers of cellular activation and blood transcriptomic profile during lupus nephritis.

ELIGIBILITY:
INCLUSION CRITERIA

For the group of 75 patients on hemodialysis

* Age ≥ 18 years,
* History of biopsy-proven lupus nephritis (all classes of lupus nephritis)

For the group of 45 patients with active lupus, not on hemodialysis

* Age ≥ 18 years,
* Biopsy-proven ACTIVE lupus nephritis

For the group of 20 healthy individuals

• Age ≥ 18 years

EXCLUSION CRITERIA

For the group of 75 patients on hemodialysis

* No written informed consent
* Past-history of kidney transplantation
* Active infection
* Active allergy (such as hay fever)
* Pregnant or breastfeeding women
* Non-affiliation to a social security regime
* Protected adults (individuals under guardianship by court order)

For the group of 45 patients with active lupus, not on hemodialysis

* No written informed consent
* Immunosuppressive therapy (except corticosteroids)
* Corticosteroids pulse before renal biopsy
* Pregnant or breastfeeding women
* Non-affiliation to a social security regime
* Protected adults (individuals under guardianship by court order)

For the group of 20 healthy individuals

* No written informed consent
* Immunosuppressive therapy (including corticosteroids)
* History of autoimmune disease
* Pregnant or breastfeeding women
* Non-affiliation to a social security regime
* Protected adults (individuals under guardianship by court order)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lupus patients on chronic haemodialysis in Ile-de-France (n=75) will be recruited for biological and clinical comparison between patients with persistent lupus activity to those with extinct lupus. These dialysis patients have been identified from the national REIN registry, which prospectively collects data for all incident patients undergoing renal replacement therapy (dialysis or kidney transplantation).
  Additionally, patients with active lupus prior to treatment and no ESRD will serve as a "positive control" group (n=45) for markers of cellular activation and blood transcriptomic profile during lupus nephritis.
  Healthy controls are required to establish reference values for assays specifically developed for the ELUDIAL study.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2022-08-11 (Actual)

PRIMARY OUTCOMES:
Nombre of patients treated by sequential haemodialysis with lupus extinction | Inclusion
  non-renal SELENA SLEDAI score < 4 and absence

CONTACTS AND LOCATIONS:
Overall Officials: Eric DAUGAS, MD PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Bichat, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Simon Q, Gaillard F, Tchen J, Bachelet D, Sacre K, Peoc'h K, Jourde-Chiche N, Daugas E, Charles N. Immune characterization of lupus nephritis patients undergoing dialysis. J Transl Autoimmun. 2025 May 2;10:100290. doi: 10.1016/j.jtauto.2025.100290. eCollection 2025 Jun. PMID 40453547